CLINICAL TRIAL: NCT00005314
Title: Behavioral Factors in Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00008338; P01HL036587 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Metabolic Syndrome X
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine and plasma samples and extracted DNA are retained
Oversight: Data Monitoring Committee: No

SUMMARY:
To elucidate the role of biobehavioral factors in the etiology, pathogenesis and course of coronary heart disease (CHD) and to use this knowledge to devise more effective prevention, treatment and rehabilitation approaches.

DETAILED DESCRIPTION:
BACKGROUND:

The integrating theme of the study is that hostility affects both behaviors and biologic functions in ways that increase the risks of developing coronary atherosclerosis or suffering an acute CHD event. Disciplines involved include psychology, internal medicine, cardiology, psychiatry, pharmacology, biostatistics, epidemiology, and molecular biology.

DESIGN NARRATIVE:

There were five subprojects in the original program project grant. Subproject 1 examined the social, behavioral and biologic concommitants of both natural and experimental interpersonal conflicts as a function of multimodal hostility assessments. Subproject 2 examined the role of hostility and social support in survival among CHD patients and attempted to identify the behavioral mediators of survival effects. Subproject 4 evaluated the effects of hostility, both alone and jointly with risk factors and social factors, on CHD incidence in over 5,000 participants in the University of North Carolina Alumni Heart Study. Subproject 5 evaluated the effects of age, smoking, lipids, and adrenergic receptors on physiologic reactivity of hostile and nonhostile men to anger induced by interpersonal challenges in the lab as well as the events of daily life. Subproject 7 extended the evaluation of anger-associated biologic reactivity in hostile and nonhostile persons by studying biobehavioral responses of 200 women employed in a real world high stress work situation; it also evaluated the impact of a stress management intervention designed to reduce anger on biobehavioral reactivity in these same employees.

The study was renewed in fiscal year (FY) 1997 to expand the primary focus on hostility to include a set of psychosocial, behavioral, and biological characteristics that increased coronary heart disease risk and appeared to cluster in certain individuals and groups, especially those low in socioeconomic status (SES). Subproject 1 examined in approximately 360 subjects the synergistic effects of SES and psychosocial risk factors such as depression, hostility, and social isolation on biological and behavioral factors suspected or known to contribute to atherogenesis. Subproject 2 evaluated the role of the central nervous system serotonin function as a potential mediator of the clustering of health-damaging psychosocial and biobehavioral characteristics in the same individuals and low SES groups. Subproject 3, the Psychosocial Risk for Cardiovascular Disease in Youth Project (PRCVDYP), used three ongoing general population studies of youth as a basis for examining the development of psychosocial risk for cardiovascular disease. The investigators hypothesized that low SES youth would exhibit, in addition to increased levels of the psychosocial and behavioral risk factors under study, increased sympathetic nervous system tone and reactivity to mental challenge, as well as decreased peripheral nervous system tone. They also hypothesized that depression, social isolation, and harsh parenting will interact with low SES to increase cardiovascular disease risk. Subproject 4 used a rat model to investigate early experience, serotonin and adult function.

The study was renewed in FY 2004 and includes three subprojects. Subproject 1 will determine the role of gene-environment interactions in the expression of psychosocial and biobehavioral risk factors for cardiovascular disease. Variants will be identified in candidate genes and chromosomal loci that are associated with the endophenotypes of hostility, personality, other psychosocial risk factors, health behaviors, and the following responses to rest and stress -- cardiovascular and neuroendocrine function, platelet activation and serotonin transporter function, circulatory inflammatory markers and the tendency of all of these characteristics to cluster in the same individuals and low socioeconomic groups. A total of 400 probands (half African American, half Caucasian, half women) and at least one sibling for each proband will be recruited for a total of 800 to 1200 subjects. Subproject 2 will explore in 400 subjects the genetics of glucose metabolism, hostility, and cardiovascular disease risk factors. Subproject 3 will examine the genetics, hostility and biology of stress in daily life in 400 probands and one sibling for every proband.

ELIGIBILITY:
We will recruit 500 probands (half African American and half Caucasian, half men and half women, and half scoring in the top and half in the bottom 20% on an established hostility scale), at least one sibling from each proband and as many parents as possible.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 694 (Actual)
Dates: Start 1986-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Manifestations of the metabolic syndrome | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Redford B Williams, M.D., Principal Investigator — Duke University

REFERENCES:
- [Background] Suarez EC, Shiller AD, Kuhn CM, Schanberg S, Williams RB Jr, Zimmermann EA. The relationship between hostility and beta-adrenergic receptor physiology in health young males. Psychosom Med. 1997 Sep-Oct;59(5):481-7. doi: 10.1097/00006842-199709000-00004. PMID 9316180
- [Background] Williams RB. The role of psychosocial factors in human disease: lessons from animal models. Acta Physiol Scand Suppl. 1997;640:100-2. PMID 9401617
- [Background] Suarez EC, Kuhn CM, Schanberg SM, Williams RB Jr, Zimmermann EA. Neuroendocrine, cardiovascular, and emotional responses of hostile men: the role of interpersonal challenge. Psychosom Med. 1998 Jan-Feb;60(1):78-88. doi: 10.1097/00006842-199801000-00017. PMID 9492244
- [Background] Muranaka M, Monou H, Suzuki J, Lane JD, Anderson NB, Kuhn CM, Schanberg SM, McCown N, Williams RB Jr. Physiological responses to catecholamine infusions in type A and type B men. Health Psychol. 1988;7 Suppl:145-63. PMID 2854049
- [Background] Barefoot JC, Peterson BL, Harrell FE Jr, Hlatky MA, Pryor DB, Haney TL, Blumenthal JA, Siegler IC, Williams RB Jr. Type A behavior and survival: a follow-up study of 1,467 patients with coronary artery disease. Am J Cardiol. 1989 Sep 1;64(8):427-32. doi: 10.1016/0002-9149(89)90416-5. PMID 2773785
- [Background] Barefoot JC, Dodge KA, Peterson BL, Dahlstrom WG, Williams RB Jr. The Cook-Medley hostility scale: item content and ability to predict survival. Psychosom Med. 1989 Jan-Feb;51(1):46-57. doi: 10.1097/00006842-198901000-00005. PMID 2928460
- [Background] Williams RB Jr. Refining the type A hypothesis: emergence of the hostility complex. Am J Cardiol. 1987 Dec 28;60(18):27J-32J. doi: 10.1016/0002-9149(87)90680-1. PMID 3321966
- [Background] Barefoot JC, Siegler IC, Nowlin JB, Peterson BL, Haney TL, Williams RB Jr. Suspiciousness, health, and mortality: a follow-up study of 500 older adults. Psychosom Med. 1987 Sep-Oct;49(5):450-7. doi: 10.1097/00006842-198709000-00002. PMID 3671634
- [Background] Suarez EC, Williams RB Jr. Situational determinants of cardiovascular and emotional reactivity in high and low hostile men. Psychosom Med. 1989 Jul-Aug;51(4):404-18. doi: 10.1097/00006842-198907000-00004. PMID 2772105
- [Background] Williams RB Jr, Barefoot JC, Haney TL, Harrell FE Jr, Blumenthal JA, Pryor DB, Peterson B. Type A behavior and angiographically documented coronary atherosclerosis in a sample of 2,289 patients. Psychosom Med. 1988 Mar-Apr;50(2):139-52. doi: 10.1097/00006842-198803000-00004. PMID 3375404
- [Background] Barefoot JC, Beckham JC, Haney TL, Siegler IC, Lipkus IM. Age differences in hostility among middle-aged and older adults. Psychol Aging. 1993 Mar;8(1):3-9. doi: 10.1037//0882-7974.8.1.3. PMID 8461112
- [Background] Barefoot JC. Keeping conflicting findings in perspective: the case of hostility and health. Mayo Clin Proc. 1993 Feb;68(2):192-3. doi: 10.1016/s0025-6196(12)60170-0. No abstract available. PMID 8423701
- [Background] Mark DB, Lam LC, Lee KL, Clapp-Channing NE, Williams RB, Pryor DB, Califf RM, Hlatky MA. Identification of patients with coronary disease at high risk for loss of employment. A prospective validation study. Circulation. 1992 Nov;86(5):1485-94. doi: 10.1161/01.cir.86.5.1485. PMID 1423962
- [Background] Barefoot JC, Beckham JC, Peterson BL, Haney TL, Williams RB Jr. Measures of neuroticism and disease status in coronary angiography patients. J Consult Clin Psychol. 1992 Feb;60(1):127-32. doi: 10.1037//0022-006x.60.1.127. PMID 1556275
- [Background] Barefoot JC, Peterson BL, Dahlstrom WG, Siegler IC, Anderson NB, Williams RB Jr. Hostility patterns and health implications: correlates of Cook-Medley Hostility Scale scores in a national survey. Health Psychol. 1991;10(1):18-24. doi: 10.1037//0278-6133.10.1.18. PMID 2026126
- [Background] Siegel WC, Hlatky MA, Mark DB, Barefoot JC, Harrell FE Jr, Pryor DB, Williams RB Jr. Effect of Type A behavior on exercise test outcome in coronary artery disease. Am J Cardiol. 1990 Jul 15;66(2):179-82. doi: 10.1016/0002-9149(90)90584-n. PMID 2196775
- [Background] Siegler IC. Paradigms in developmental health psychology--from theory to application: introduction to a special issue. J Gerontol. 1990 Jul;45(4):P113-5. doi: 10.1093/geronj/45.4.p113. PMID 2365967
- [Background] Siegler IC, Peterson BL, Barefoot JC, Harvin SH, Dahlstrom WG, Kaplan BH, Costa PT Jr, Williams RB Jr. Using college alumni populations in epidemiologic research: the UNC Alumni Heart Study. J Clin Epidemiol. 1992 Nov;45(11):1243-50. doi: 10.1016/0895-4356(92)90165-j. PMID 1432005
- [Background] Siegler IC, Peterson BL, Barefoot JC, Williams RB. Hostility during late adolescence predicts coronary risk factors at mid-life. Am J Epidemiol. 1992 Jul 15;136(2):146-54. doi: 10.1093/oxfordjournals.aje.a116481. PMID 1415138
- [Background] Williams RB Jr, Suarez EC, Kuhn CM, Zimmerman EA, Schanberg SM. Biobehavioral basis of coronary-prone behavior in middle-aged men. Part I: Evidence for chronic SNS activation in Type As. Psychosom Med. 1991 Sep-Oct;53(5):517-27. doi: 10.1097/00006842-199109000-00003. PMID 1661901
- [Background] Suarez EC, Williams RB Jr, Kuhn CM, Zimmerman EH, Schanberg SM. Biobehavioral basis of coronary-prone behavior in middle-age men. Part II: Serum cholesterol, the Type A behavior pattern, and hostility as interactive modulators of physiological reactivity. Psychosom Med. 1991 Sep-Oct;53(5):528-37. doi: 10.1097/00006842-199109000-00004. PMID 1758939
- [Background] Suarez EC, Harlan E, Peoples MC, Williams RB Jr. Cardiovascular and emotional responses in women: the role of hostility and harassment. Health Psychol. 1993 Nov;12(6):459-68. doi: 10.1037//0278-6133.12.6.459. PMID 8293729
- [Background] Siegler IC, Zonderman AB, Barefoot JC, Williams RB Jr, Costa PT Jr, McCrae RR. Predicting personality in adulthood from college MMPI scores: implications for follow-up studies in psychosomatic medicine. Psychosom Med. 1990 Nov-Dec;52(6):644-52. doi: 10.1097/00006842-199011000-00006. PMID 2287703
- [Background] Suarez EC, Williams RB Jr. The relationships between dimensions of hostility and cardiovascular reactivity as a function of task characteristics. Psychosom Med. 1990 Sep-Oct;52(5):558-70. doi: 10.1097/00006842-199009000-00008. PMID 2247561
- [Background] Williams RB, Barefoot JC, Blumenthal JA, Helms MJ, Luecken L, Pieper CF, Siegler IC, Suarez EC. Psychosocial correlates of job strain in a sample of working women. Arch Gen Psychiatry. 1997 Jun;54(6):543-8. doi: 10.1001/archpsyc.1997.01830180061007. PMID 9193195
- [Background] Siegler HC, Blumenthal JA, Barefoot JC, Peterson BL, Saunders WB, Dahlstrom WG, Costa PT Jr, Suarez EC, Helms MJ, Maynard KE, Williams RB. Personality factors differentially predict exercise behavior in men and women. Womens Health. 1997 Spring;3(1):61-70. PMID 9106371
- [Background] Von Dras DD, Siegler IC. Stability in extraversion and aspects of social support at midlife. J Pers Soc Psychol. 1997 Jan;72(1):233-41. doi: 10.1037//0022-3514.72.1.233. PMID 9008383
- [Background] Haney TL, Maynard KE, Houseworth SJ, Scherwitz LW, Williams RB, Barefoot JC. Interpersonal Hostility Assessment Technique: description and validation against the criterion of coronary artery disease. J Pers Assess. 1996 Apr;66(2):386-401. doi: 10.1207/s15327752jpa6602_16. PMID 8869579
- [Background] Harrell FE Jr, Lee KL, Mark DB. Multivariable prognostic models: issues in developing models, evaluating assumptions and adequacy, and measuring and reducing errors. Stat Med. 1996 Feb 28;15(4):361-87. doi: 10.1002/(SICI)1097-0258(19960229)15:43.0.CO;2-4. PMID 8668867
- [Background] Dawson DV, Siegler IC. Approaches to the nonparametric analysis of limited longitudinal data sets. Exp Aging Res. 1996 Jan-Mar;22(1):33-57. doi: 10.1080/03610739608253996. PMID 8665986
- [Background] Barefoot JC, Larsen S, von der Lieth L, Schroll M. Hostility, incidence of acute myocardial infarction, and mortality in a sample of older Danish men and women. Am J Epidemiol. 1995 Sep 1;142(5):477-84. doi: 10.1093/oxfordjournals.aje.a117663. PMID 7677126
- [Background] Lipkus IM, Siegler IC. Do comparative self-appraisals during young adulthood predict adult personality? Psychol Aging. 1995 Jun;10(2):229-37. doi: 10.1037//0882-7974.10.2.229. PMID 7662182
- [Background] Anderson NB, Armstead CA. Toward understanding the association of socioeconomic status and health: a new challenge for the biopsychosocial approach. Psychosom Med. 1995 May-Jun;57(3):213-25. doi: 10.1097/00006842-199505000-00003. PMID 7652122
- [Background] Siegler IC, Feaganes JR, Rimer BK. Predictors of adoption of mammography in women under age 50. Health Psychol. 1995 May;14(3):274-8. doi: 10.1037//0278-6133.14.3.274. PMID 7641669
- [Background] Williams RB. Neurobiology, cellular and molecular biology, and psychosomatic medicine. Psychosom Med. 1994 Jul-Aug;56(4):308-15. doi: 10.1097/00006842-199407000-00006. No abstract available. PMID 7972613
- [Background] Barefoot JC, Patterson JC, Haney TL, Cayton TG, Hickman JR Jr, Williams RB. Hostility in asymptomatic men with angiographically confirmed coronary artery disease. Am J Cardiol. 1994 Sep 1;74(5):439-42. doi: 10.1016/0002-9149(94)90899-0. PMID 8059722
- [Background] Lipkus IM, Barefoot JC, Williams RB, Siegler IC. Personality measures as predictors of smoking initiation and cessation in the UNC Alumni Heart Study. Health Psychol. 1994 Mar;13(2):149-55. doi: 10.1037//0278-6133.13.2.149. PMID 8020458
- [Background] Von Dras DD, Siegler IC, Williams RB, Clapp-Channing N, Haney TL, Mark DB. Surrogate assessment of coronary artery disease patients' functional capacity. Soc Sci Med. 1997 May;44(10):1491-502. doi: 10.1016/s0277-9536(96)00269-9. PMID 9160439
- [Background] Von Dras DD, Williams RB, Kaplan BH, Siegler IC. Correlates of perceived social support and equality of interpersonal relationships at mid-life. Int J Aging Hum Dev. 1996;43(3):199-217. doi: 10.2190/M0GP-7R75-AQJ6-Q17H. PMID 9031005
- [Background] Hlatky MA, Lam LC, Lee KL, Clapp-Channing NE, Williams RB, Pryor DB, Califf RM, Mark DB. Job strain and the prevalence and outcome of coronary artery disease. Circulation. 1995 Aug 1;92(3):327-33. doi: 10.1161/01.cir.92.3.327. PMID 7634445
- [Background] Barefoot JC, Helms MJ, Mark DB, Blumenthal JA, Califf RM, Haney TL, O'Connor CM, Siegler IC, Williams RB. Depression and long-term mortality risk in patients with coronary artery disease. Am J Cardiol. 1996 Sep 15;78(6):613-7. doi: 10.1016/s0002-9149(96)00380-3. PMID 8831391
- [Background] Lane JD, Pieper CF, Barefoot JC, Williams RB Jr, Siegler IC. Caffeine and cholesterol: interactions with hostility. Psychosom Med. 1994 May-Jun;56(3):260-6. doi: 10.1097/00006842-199405000-00013. PMID 8084973
- [Background] Lipkus IM, Barefoot JC, Feaganes J, Williams RB, Siegler IC. A short MMPI scale to identify people likely to begin smoking. J Pers Assess. 1994 Apr;62(2):213-22. doi: 10.1207/s15327752jpa6202_4. PMID 8189332
- [Background] Brummett BH, Barefoot JC, Feaganes JR, Yen S, Bosworth HB, Williams RB, Siegler IC. Hostility in marital dyads: associations with depressive symptoms. J Behav Med. 2000 Feb;23(1):95-105. doi: 10.1023/a:1005424405056. PMID 10749013
- [Background] Bosworth HB, Siegler IC, Brummett BH, Barefoot JC, Williams RB, Clapp-Channing NE, Mark DB. The association between self-rated health and mortality in a well-characterized sample of coronary artery disease patients. Med Care. 1999 Dec;37(12):1226-36. doi: 10.1097/00005650-199912000-00006. PMID 10599604
- [Background] Brummett BH, Maynard KE, Babyak MA, Haney TL, Siegler IC, Helms MJ, Barefoot JC. Measures of hostility as predictors of facial affect during social interaction: evidence for construct validity. Ann Behav Med. 1998 Summer;20(3):168-73. doi: 10.1007/BF02884957. PMID 9989323
- [Background] Brummett BH, Babyak MA, Barefoot JC, Bosworth HB, Clapp-Channing NE, Siegler IC, Williams RB Jr, Mark DB. Social support and hostility as predictors of depressive symptoms in cardiac patients one month after hospitalization: a prospective study. Psychosom Med. 1998 Nov-Dec;60(6):707-13. doi: 10.1097/00006842-199811000-00008. PMID 9847029
- [Background] Barefoot JC, Heitmann BL, Helms MJ, Williams RB, Surwit RS, Siegler IC. Symptoms of depression and changes in body weight from adolescence to mid-life. Int J Obes Relat Metab Disord. 1998 Jul;22(7):688-94. doi: 10.1038/sj.ijo.0800647. PMID 9705031
- [Background] Williams RB. The mind, the body, health, and disease. What do we know, what should we do? N C Med J. 1998 May-Jun;59(3):172-4. No abstract available. PMID 9610159
- [Background] Luecken LJ, Suarez EC, Kuhn CM, Barefoot JC, Blumenthal JA, Siegler IC, Williams RB. Stress in employed women: impact of marital status and children at home on neurohormone output and home strain. Psychosom Med. 1997 Jul-Aug;59(4):352-9. doi: 10.1097/00006842-199707000-00003. PMID 9251153
- [Background] Bosworth HB, Siegler IC, Olsen MK, Brummett BH, Barefoot JC, Williams RB, Clapp-Channing NE, Mark DB. Social support and quality of life in patients with coronary artery disease. Qual Life Res. 2000;9(7):829-39. doi: 10.1023/a:1008960308011. PMID 11297025
- [Background] Williams RB, Marchuk DA, Gadde KM, Barefoot JC, Grichnik K, Helms MJ, Kuhn CM, Lewis JG, Schanberg SM, Stafford-Smith M, Suarez EC, Clary GL, Svenson IK, Siegler IC. Central nervous system serotonin function and cardiovascular responses to stress. Psychosom Med. 2001 Mar-Apr;63(2):300-5. doi: 10.1097/00006842-200103000-00016. PMID 11292279
- [Background] Brummett BH, Barefoot JC, Siegler IC, Clapp-Channing NE, Lytle BL, Bosworth HB, Williams RB Jr, Mark DB. Characteristics of socially isolated patients with coronary artery disease who are at elevated risk for mortality. Psychosom Med. 2001 Mar-Apr;63(2):267-72. doi: 10.1097/00006842-200103000-00010. PMID 11292274
- [Background] Williams RB. Hostility and heart disease: Williams et al. (1980). Adv Mind Body Med. 2001 Winter;17(1):52-5. No abstract available. PMID 11270067
- [Background] Barefoot JC, Brummett BH, Helms MJ, Mark DB, Siegler IC, Williams RB. Depressive symptoms and survival of patients with coronary artery disease. Psychosom Med. 2000 Nov-Dec;62(6):790-5. doi: 10.1097/00006842-200011000-00008. PMID 11138998
- [Background] Brummett BH, Maynard KE, Haney TL, Siegler IC, Barefoot JC. Reliability of interview-assessed hostility ratings across mode of assessment and time. J Pers Assess. 2000 Oct;75(2):225-36. doi: 10.1207/S15327752JPA7502_4. PMID 11020141
- [Background] Barefoot JC, Brummett BH, Clapp-Channing NE, Siegler IC, Vitaliano PP, Williams RB, Mark DB. Moderators of the effect of social support on depressive symptoms in cardiac patients. Am J Cardiol. 2000 Aug 15;86(4):438-42. doi: 10.1016/s0002-9149(00)00961-9. PMID 10946039
- [Background] Bosworth HB, Siegler IC, Brummett BH, Barefoot JC, Williams RB, Vitaliano PP, Clapp-Channing N, Lytle BL, Mark DB. The relationship between self-rated health and health status among coronary artery patients. J Aging Health. 1999 Nov;11(4):565-84. doi: 10.1177/089826439901100405. PMID 10848078
- [Background] Von Dras DD, Siegler IC, Barefoot JC, Williams RB, Mark DB. Coronary catherization patient and wife's perceptions of social support: effects due to characteristics of recipient, provider, and their interaction. Int J Aging Hum Dev. 2000;50(2):97-125. doi: 10.2190/CU9W-0XKW-R4AN-G1TD. PMID 10791611
- [Background] Barefoot JC, Mortensen EL, Helms MJ, Avlund K, Schroll M. A longitudinal study of gender differences in depressive symptoms from age 50 to 80. Psychol Aging. 2001 Jun;16(2):342-5. doi: 10.1037//0882-7974.16.2.342. PMID 11405320
- [Background] Siegler IC, Bastian LA, Steffens DC, Bosworth HB, Costa PT. Behavioral medicine and aging. J Consult Clin Psychol. 2002 Jun;70(3):843-51. doi: 10.1037//0022-006x.70.3.843. PMID 12090387
- [Background] Brummett BH, Babyak MA, Mark DC, Williams RB, Siegler IC, Clapp-Channing N, Barefoot JC. Predictors of smoking cessation in patients with a diagnosis of coronary artery disease. J Cardiopulm Rehabil. 2002 May-Jun;22(3):143-7. doi: 10.1097/00008483-200205000-00003. PMID 12042680
- [Background] Williams RB, Marchuk DA, Gadde KM, Barefoot JC, Grichnik K, Helms MJ, Kuhn CM, Lewis JG, Schanberg SM, Stafford-Smith M, Suarez EC, Clary GL, Svenson IK, Siegler IC. Serotonin-related gene polymorphisms and central nervous system serotonin function. Neuropsychopharmacology. 2003 Mar;28(3):533-41. doi: 10.1038/sj.npp.1300054. Epub 2002 Aug 29. PMID 12629534
- [Background] Williams RB, Schneiderman N. Resolved: psychosocial interventions can improve clinical outcomes in organic disease (pro). Psychosom Med. 2002 Jul-Aug;64(4):552-7. doi: 10.1097/01.psy.0000023410.02546.5d. No abstract available. PMID 12140342
- [Background] Surwit RS, Williams RB, Siegler IC, Lane JD, Helms M, Applegate KL, Zucker N, Feinglos MN, McCaskill CM, Barefoot JC. Hostility, race, and glucose metabolism in nondiabetic individuals. Diabetes Care. 2002 May;25(5):835-9. doi: 10.2337/diacare.25.5.835. PMID 11978677
- [Background] Williams RB, Barefoot JC, Schneiderman N. Psychosocial risk factors for cardiovascular disease: more than one culprit at work. JAMA. 2003 Oct 22;290(16):2190-2. doi: 10.1001/jama.290.16.2190. No abstract available. PMID 14570955
- [Background] Williams RB. Invited commentary: socioeconomic status, hostility, and health behaviors--does it matter which comes first? Am J Epidemiol. 2003 Oct 15;158(8):743-6. doi: 10.1093/aje/kwg205. No abstract available. PMID 14561663
- [Background] Burroughs AR, Visscher WA, Haney TL, Efland JR, Barefoot JC, Williams RB Jr, Siegler IC. Community recruitment process by race, gender, and SES gradient: lessons learned from the Community Health and Stress Evaluation (CHASE) Study experience. J Community Health. 2003 Dec;28(6):421-37. doi: 10.1023/a:1026029723762. PMID 14620965
- [Background] Siegler IC, Costa PT, Brummett BH, Helms MJ, Barefoot JC, Williams RB, Dahlstrom WG, Kaplan BH, Vitaliano PP, Nichaman MZ, Day RS, Rimer BK. Patterns of change in hostility from college to midlife in the UNC Alumni Heart Study predict high-risk status. Psychosom Med. 2003 Sep-Oct;65(5):738-45. doi: 10.1097/01.psy.0000088583.25140.9c. PMID 14508014
- [Background] Brummett BH, Babyak MA, Siegler IC, Mark DB, Williams RB, Barefoot JC. Effect of smoking and sedentary behavior on the association between depressive symptoms and mortality from coronary heart disease. Am J Cardiol. 2003 Sep 1;92(5):529-32. doi: 10.1016/s0002-9149(03)00719-7. PMID 12943871
- [Background] Brummett BH, Barefoot JC, Vitaliano PP, Siegler IC. Associations among social support, income, and symptoms of depression in an educated sample: the UNC Alumni Heart Study. Int J Behav Med. 2003;10(3):239-50. doi: 10.1207/s15327558ijbm1003_04. PMID 14525719
- [Background] Boyle SH, Williams RB, Mark DB, Brummett BH, Siegler IC, Helms MJ, Barefoot JC. Hostility as a predictor of survival in patients with coronary artery disease. Psychosom Med. 2004 Sep-Oct;66(5):629-32. doi: 10.1097/01.psy.0000138122.93942.4a. PMID 15385683
- [Background] Williams RB. Treating depression after myocardial infarction: can selecting patients on the basis of genetic susceptibility improve psychiatric and medical outcomes? Am Heart J. 2005 Oct;150(4):617-9. doi: 10.1016/j.ahj.2005.04.028. No abstract available. PMID 16209955
- [Background] Zhang X, Gainetdinov RR, Beaulieu JM, Sotnikova TD, Burch LH, Williams RB, Schwartz DA, Krishnan KR, Caron MG. Loss-of-function mutation in tryptophan hydroxylase-2 identified in unipolar major depression. Neuron. 2005 Jan 6;45(1):11-6. doi: 10.1016/j.neuron.2004.12.014. PMID 15629698
- [Background] Brummett BH, Boyle SH, Siegler IC, Williams RB, Mark DB, Barefoot JC. Ratings of positive and depressive emotion as predictors of mortality in coronary patients. Int J Cardiol. 2005 Apr 20;100(2):213-6. doi: 10.1016/j.ijcard.2004.06.016. PMID 15823627
- [Background] Brummett BH, Mark DB, Siegler IC, Williams RB, Babyak MA, Clapp-Channing NE, Barefoot JC. Perceived social support as a predictor of mortality in coronary patients: effects of smoking, sedentary behavior, and depressive symptoms. Psychosom Med. 2005 Jan-Feb;67(1):40-5. doi: 10.1097/01.psy.0000149257.74854.b7. PMID 15673622
- [Background] Boyle SH, Williams RB, Mark DB, Brummett BH, Siegler IC, Barefoot JC. Hostility, age, and mortality in a sample of cardiac patients. Am J Cardiol. 2005 Jul 1;96(1):64-6. doi: 10.1016/j.amjcard.2005.02.046. PMID 15979435